CLINICAL TRIAL: NCT01589380
Title: Safety and Efficacy of Angiotensin Receptor Blocker, Fimasartan, on Patients With Aortic Stenosis
Brief Title: A Randomized Trial of Angiotensin Receptor bLocker,Fimasartan, in Aortic Stenosis (ALFA Trial)
Acronym: ALFA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry); Seoul National University Bundang Hospital (Other); Severance Hospital (Other); Korea University Anam Hospital (Other); Korea University Guro Hospital (Other); Chonnam National University Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yong-Jin Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCT16453143
Record Dates: First submitted 2012-04-29; First posted 2012-05-01 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Critical Stenosis of Aortic Valve
Keywords: Aortic stenosis; Exercise performance; cardiopulmonary exercise test; fimasartan
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — fimasartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Arm (Placebo Comparator): Placebo: Capsule that is containing lactate hydrate, identically appearing with fimasartan will be administered to patient in placebo group, once daily. Same placebo drug which was used in phase 3 clinical trial of fimasartan will be provided by Boryoung Phamaceutical company. Dose titration will be done with same criteria of fimasartan group. 30mg form and 60 mg form of placebo will be identical in its morphology.
  Interventions: Drug: Placebo
- Fimasartan (Active Comparator): Fimasartan, Initial dose will be started with 30mg per day. At 12 months follow-up after the enrollment, dose titration up to 60 mg per day will be made with target blood pressure of 120/80.
  Dose escalization from 30mg/day to 60mg/day will be performed in the case of follow-up systolic blood pressure is over 120. If the follow-up systolic blood pressure is less than 120, initial dose of 30mg/day will be maintained throughout the study duration. If hypotension (BP < 90/60) is developed, the study medication will be discontinued and the patient will be included safety outcome analysis and intention to treat analysis. Per protocol analysis will be also performed. The dose of placebo will be adjusted identically, according to the blood pressure criteria of fimasartan.
  Interventions: Drug: Fimasartan

INTERVENTIONS:
Drug: Fimasartan — Fimasartan, Initial dose will be started with 30mg per day. At 12 months follow-up after the enrollment, dose titration up to 60 mg per day will be made with target blood pressure of 120/80.
  Dose escalization from 30mg/day to 60mg/day will be performed in the case of follow-up systolic blood pressure is over 120. If the follow-up systolic blood pressure is less than 120, initial dose of 30mg/day will be maintained throughout the study duration. If hypotension (BP < 90/60) is developed, the study medication will be discontinued and the patient will be included safety outcome analysis and intention to treat analysis. Per protocol analysis will be also performed. The dose of placebo will be adjusted identically, according to the blood pressure criteria of fimasartan.
  Other Names: Fimasartan (BR-A-657; CAS : 247257-48-3; Kanarb)
  Arms: Fimasartan
Drug: Placebo — Placebo was used in phase 3 clinical trial of fimasartan (NCT00922480, NCT01135212, and NCT01258673). The same placebo, which is manufactures at Boryoung pharmaceutical company, will be used in this trial. After enrollment and randomization, placebo will be administered one capsule once daily in placebo group.
  Other Names: Lactose Hydrate
  Arms: Placebo Arm

SUMMARY:
We hypothesized that fimasartan, a new generation ARBs, would improve exercise capacity and decrease the rate of progression of AS by modifying hemodynamic factors and reducing adverse LV remodeling favorably in patients with asymptomatic moderate to severe AS.

DETAILED DESCRIPTION:
Aortic stenosis (AS) is common valvular disorder, affecting 2% to 4% of adults older than 65 years. It is gradually but constantly progressive disease whit a long asymptomatic phase, but once symptoms develop, the prognosis is poor.

Currently, treatment strategy is focused mainly to watchful monitoring and judicious timing of aortic valve replacement (AVR). However, not all patients are proper candidate of corrective surgery and the needs of development of medical treatment are increasing. Various mechanisms have been suggested in progression of AS and recent observational studies suggested not only mechanical stress of "wear and tear" but also active inflammatory process likewise atherosclerosis may contribute the progression of AS. Through clinical descriptive studies, atherosclerotic risk factors, such as hypertension, diabetes mellitus, dyslipidemia, obesity, smoking, and metabolic syndrome have been known to facilitate the progression of AS.

The renin-angiotensin system (RAS) is activated at an early stage of AS, promoting developemtnt of left ventricular hypertrophy (LVH), myocardial fibrosis, and diastolic dysfunction. Lipid lowering therapy and RAS blockade have emerged potential medical treatment to slow the progression of AS, however, many clinical trials did not show consistent beneficial effect of statins.8-10 RAS blockers are perceived as being relative contraindication due to concerns about increasing pressure gradient. However, patients with AS tolerate RAS blocker well on initiation and the use of angiotensin converting enzyme (ACE) inhibitors appears to confer long term survival benefit on patients considered to have a contraindication including AS.Pressure overload of LV, activation of RAS, and subsequent adverse LV remodeling, myocardial fibrosis, and LV dysfunction may potential therapeutic target to retard the progression of AS and to improve exercise capacity, and even long-term outcomes. RAS blocker including ACEI or angiotensin receptor blockers (ARBs) have been known to improve exercise capacity and long term outcome in patient with hypertension, congestive heart failure, or myocardial infarction.

We hypothesized that fimasartan, a new generation ARBs, would improve exercise capacity and decrease the rate of progression of AS by modifying hemodynamic factors and reducing adverse LV remodeling favorably in patients with asymptomatic moderate to severe AS.

Prospective, double-blinded, randomized clinical trial with enrollment of normotensive or hypertensive patients of age 20 to 75 who require echocardiography for a clinical indication, which typically consists of known aortic stenosis or presence of cardiac murmur. Moderate to severe aortic stenosis will be defined as a continuous wave Doppler determined peak aortic valve jet velocity of 3.0 - 4.5 m/s or mean pressure gradient of 25 - 49 mmHg, or aortic valve area of 0.76 - 1.5 cm2. Patients meeting inclusion criteria without any exclusion criteria will be randomized 1:1 to angiotensin receptor blocker, Fimasartan, or placebo. After 1-year enrollment period, all patients will be followed for 1 year. Cardiopulmonary exercise test will be performed at baseline enrollment period, and at the end of follow-up. Echocardiographic evaluation will be performed at regular interval of baseline and 6 months interval until the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age: 20-75 years
* Moderate to severe aortic stenosis defined as a continuous wave Doppler determined peak aortic valve jet velocity of 3.0 - 4.5 m/s, mean pressure gradient of 25 - 49 mmHg, or aortic valve area of 0.76 - 1.5 cm2.
* Asymptomatic aortic stenosis patients, Stationary or minimum dyspnea on exertion (NYHA Fc ≤ I or II) will be included.
* Patients who were prescribed ACEI or ARBs for treatment of hypertension will be enrolled after 2 weeks wash-out period.
* SBP 120-140 mmHg with or without medication regardless of presence of hypertension or not.
* Patients with BP > 140/90 mmHg with or without medication will be included after their BP is controlled with anti-hypertensive medication other than ACEI/ARBs.
* Patients who are able to perform appropriate cardiopulmonary exercise test with treadmill.
* The patient agrees to the study protocol and the schedule of clinical, cardiopulmonary exercise test, and echocardiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Symptomatic aortic stenosis: presence of exertional dyspnea (≥ NYHA Fc III), angina or syncope
* Very severe aortic stenosis regardless of presence of symptoms. It was defined as a critical stenosis in the aortic valve area ≤ 0.75 cm2 accompanied by a peak aortic jet velocity ≥4.5 m/s or a mean transaortic pressure gradient ≥50 mm Hg on Doppler echocardiography.
* Uncontrolled HTN (SBP > 160 or DBP >100) without ACEI or ARBs during 2-weeks wash out period in patients who were prescribed ACEI or ARBs for treatment of hypertension.
* Patients with known history of coronary artery disease including myocardial infarction, regardless of the treatment (medication only, percutaneous coronary intervention, or coronary artery bypass grafting).
* Planned cardiac surgery or planned major non-cardiac surgery within the study period.
* Stroke or resuscitated sudden death in the past 6 months.
* Chronic disease requiring treatment with oral, intravenous, or intra-articular corticosteroids (use of topical, or nasal corticosteroids is permissible).
* Untreated hyperthyroidism or hypothyroidism with TSH levels more than 2 times upper limit of normal.
* A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer.
* Female of child-bearing potential who do not use adequate contraception and women who are pregnant or breast-feeding.
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* Evidence of congestive heart failure, or left ventricular ejection fraction < 50%.
* Significant renal disease manifested by serum creatinine > 2.0mg/dL
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal).
* Documented bilateral renal artery stenosis or known contraindication of ACEI or ARBs
* History of chronic obstructive pulmonary disease or asthma manifested by acute aggravation of COPD in the past 6 months, or currently taking bronchodilators including long-acting beta2 agonist, anticholinergics, or inhaled steroids.
* Other valvular disease : Moderate or severe mitral regurgitation or mitral stenosis, Moderate or severe aortic regurgitation
* Patients who are unable to perform cardiopulmonary exercise test.
* Unwillingness or inability to comply with the procedures described in this protocol.
* Patient who have been diagnosed with galactose intolerance, lactase deficiency, malabsorption of glucose or galactose which is main ingredient of placebo.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-05 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change of VmaxO2 in Cardiopulmonary Exercise Test | Baseline and 1 year
  Change of VmaxO2 from baseline to 1 year follow-up. VmaxO2 is defined as the highest oxygen uptake, averaged over 5 consecutive breaths, during the last minute of symptom-limited cardiopulmonary exercise test. For each patient, the change in VamxO2 is calculated as (VmaxO2 at 1 year follow-up) - (VmaxO2 at baseline)

SECONDARY OUTCOMES:
Change of peak aortic jet velocity in echocardiography | Baseline and 1 year
  Change of peak aortic jet velocity which defined as (peak aortic jet velocity at 1 year follow-up) - (peak aortic jet velocity at baseline) on Doppler echocardiography.
Change of mean pressure gradient across aortic valve | Baseline and 1 year
  Change of mean pressure gradient which will be measured in echocardiography from baseline to study end.
Diastolic function - LA area (cm2), E/E' value | Baseline and 1 year
  Change of LA area (cm2), E/E' value measured with Doppler echocardiography from baseline to study end
Left ventricular mass index (LVMI) | Baseline and 1 year
  Change of LVMI from baseline to study end.
Development of aortic stenosis symptoms | Baseline and 1 year
  Development of aortic stenosis symptoms angina, dyspnea, or syncope
Admission for heart failure | Baseline and 1 year
  During 1 year follow-up, admission due to congestiv eheart failure will be evaluated as secondary clinical outcome.
Development of left ventricular dysfunction (LVEF <50%) | Baseline and 1 year
  During follow-up, the development of LV dysfunction in echocardiography will be evaluated.
Aortic valve surgery | Baseline and 1 year
  During 1 year follow-up, the incidence of aortic valver surgery will be evaluated.
Cardiac death including Sudden cardiac death | Baseline and 1 year
  Cardiac death
All-cause death | Baseline and 1 year
  All-cause mortality
Composite Clinical Endpoint | Baseline and 1 year
  Composite Endpoint which is consist of following:
  Development of symptom of aortic stenosis: angina, dyspnea, or syncope Admission for heart failure Development of left ventricular dysfunction (LVEF <50%) Aortic valve surgery Cardiac death including Sudden cardiac death (will be collected separately) All-cause death Individual components of composite endpoint will be investigated separately also
6-minutes walk distance | Baseline and 1 year
  6-minutes walk distance from baseline to 1 year follow-up. For each patient, the change in 6-minutes walk distance is calculated as (6-minutes walk distance at 1 year follow-up) - (6-minutes walk distance at baseline)
Safety Endpoint | Baseline and 1 year
  1. Development of symptomatic hypotension (dizziness, orthostatic hypotension with BP < 90/60)
  2. Development of overt azotemia (serum creatinine > 2.0mg/dL)
  3. Intolerance or development of other adverse drug reactions related with study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Jin Kim, MD,PhD, Study Chair — Seoul National University Hospital; Seung-Pyo Lee, MD, Study Director — Seoul National University Hospital; Joo Myung Lee, MD, Study Director — Seoul National University Hospital; Sung-Ji Park, MD,PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine; Goo-Yeong Cho, MD,PhD, Principal Investigator — Seoul National University Bundang Hospital; Hyung-Kwan Kim, MD, PhD, Study Director — Seoul National University Hospital; Seong-Mi Park, Principal Investigator — Korea University Anam Hospital; Seong Woo Han, Principal Investigator — Korea University Guro Hospital; Kye Hun Kim, Principal Investigator — Chonnam University Hospital; Geu-Ru Hong, Principal Investigator — Yonsei University Hospital
Locations (7):
- South Korea (7):
  - Chonnam University Hospital, Gwangju, Gwangju
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, Seoul
  - Korea University Anam Hospital, Seoul, Seoul
  - Korea University Guro Hospital, Seoul, Seoul
  - Yonsei University Hospital, Seoul, Seoul